CLINICAL TRIAL: NCT01746797
Title: Symptom Tracking in Women With a History of Depression Going Through Infertility Treatment.
Brief Title: Symptom Tracking in Assisted Reproductive Technologies
Acronym: START
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Marlene P. Freeman, MD, Director of Clinical Services at the Center for Women's Mental Health, Massachusetts General Hospital
Other Study IDs: 2012P001637
Record Dates: First submitted 2012-12-07; First posted 2012-12-11 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Depression Relapse in Women Undergoing Fertility Treatment
Keywords: infertility; depression; IVF; IUI; fertility treatment
MeSH Terms: conditions — Infertility; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — samples obtained with permission from participant and stored for future proteomic research

GROUPS / COHORTS (2):
- Women currently taking antidepressants: Women who have selected to stay on antidepressant medication while undergoing infertility treatment.
- Women not on antidepressants: Women who decided to discontinue their antidepressants while undergoing fertility treatments.

SUMMARY:
This study assesses risk factors for depressive relapse in women undergoing fertility treatment with histories of major depressive disorder (MDD) or bipolar disorder. The study is focused on the acute risk factors of depressive relapse.

The investigators hypothesize that risk for depressive relapse will be greater among women who stop antidepressants compared to those who continue treatment with these agents.

DETAILED DESCRIPTION:
This study hopes to address the following aims:

Specific Aim #1: To delineate the relative risk of relapse in women undergoing IVF, IUI, or other infertility treatments who discontinue antidepressant therapy for depression, compared to those who maintain treatment with these agents.

Hypothesis: Risk for depressive relapse will be greater among women who stop antidepressants compared to those who continue treatment with these agents.

Specific Aim #2: To identify predictors of depressive relapse among women receiving IVF, IUI, or other infertility treatments

Hypothesis: Relapse rates will be greater among those who have: 1) histories of more recurrent depressive illness, 2) longer duration of attempt to conceive, and 3) a lower degree of perceived support from respective partners.

Specific Aim #3 (exploratory): To describe the trajectory of depressive symptoms in women with histories of depression across the course of IVF, IUI, or other treatments.

Hypothesis: Specific phases of the IVF cycle will have differential effects on the burden of depressive symptoms. Specifically, these phases include: 1) the phase prior to egg retrieval, 2) the phase after embryo transfer while a woman waits for the pregnancy test or her menstrual period, and 3) the phase after the experience of a negative pregnancy test (when applicable) following an IVF cycle. We seek to characterize factors associated both with vulnerability to more depressive symptoms and to resilience in the context of the different phases of IVF treatment.

Specific Aim #4 (exploratory): To identify biological markers of stress, including HPA axis dysregulation and inflammation associated with depressive relapse, during IVF, IUI, or other infertility treatments

Hypothesis: Hypothalamic-pituitary-adrenal (HPA) axis dysregulation, evidenced by increases in diurnal salivary cortisol patterns and markers of inflammation, will be associated with higher

ELIGIBILITY:
Inclusion Criteria:

* Have a history of a MDE or bipolar disorder prior to starting fertility treatment.
* Have received consultation around infertility treatment and plan to start fertility treatment.

Exclusion Criteria:

* Use of corticosteroids within 1 month of enrollment.
* Presence of any endocrine or autoimmune disorder, other than hypothyroidism well-treated for at least 6 months.
* Current episode of depression or mania.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will include 60 women 18 years and older with histories of depression or bipolar disorder who are planning infertility treatment, specifically in utero insemination (IUI) or in vitro fertilization (IVF).
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2012-10; Primary Completion 2016-06 (Actual); Study Completion 2018-01-16 (Actual)

PRIMARY OUTCOMES:
Depression relapse | six months

CONTACTS AND LOCATIONS:
Overall Officials: Marlene F Freeman, MD, Principal Investigator — Massachusetts General Hospital; Lee S Cohen, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States